CLINICAL TRIAL: NCT04530227
Title: A Pilot Study of Camrelizumab With Chemotherapy in Adults With Medically Inoperable Early Stage Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Camrelizumab With Chemotherapy in Adults With Medically Inoperable Early Stage NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-NSCLC-II-007
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-08

CONDITIONS: Early Stage Non-small Cell Lung Cancer
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death-ligand 1 (PD-L1, PDL1)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — camrelizumab; Pemetrexed; 130-nm albumin-bound paclitaxel; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab combined with chemotherapy (Experimental): Participants receive camrelizumab 200 mg by intravenous (IV) infusion prior to chemotherapy on Day 1 of each 21-day cycle for up to 18 cycles PLUS Investigator's choice of chemotherapy.
  Interventions:
  Biological: Camrelizumab
  Interventions: Drug: Biological: Camrelizumab; Drug: Pemetrexed; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Biological: Camrelizumab — PD-1
  Other Names: SHR-1210
Drug: Pemetrexed — chemotherapy
  Other Names: Pemetrexed Disodium
Drug: Nab-paclitaxel — chemotherapy
  Other Names: Paclitaxel for Injection（Albumin Bound）

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Camrelizumab plus chemotherapy in the treatment of adult participants with medically inoperable Stage I or IIA non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This trial will evaluate the safety and efficacy of camrelizumab in combination with chemotherapy, followed by camrelizumab alone after 4-6 cycles of combination in participants with medically inoperable stage I or IIA non-small cell lung cancer (NSCLC). The primary objective of this pilot study is to determine the Camrelizumab plus chemotherapy improves progression-free survival (PFS) . All the efficacy and safety are assessed by investigator : 1) response rate (ORR), 2) disease control rate (DCR); 3) overall survival (OS), 4) PFS rate of 1-year, 2-year, and 5-year; and 5) OS rate of 1-year, 2-year, and 5-year.

Explore objective is potential biomarker associated with efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years, male and female are not limited;
2. Patients with ECOG score of 0-1;
3. Life expectancy ≥12 weeks;
4. Patients must have histologically- or cytologically-documented NSCLC (according to 2015 WHO Classification);
5. Patients with stage I - IIA (T1-T2bN0M0, tumor size ≤ 50mm) confirmed by radiographic；and medical inoperable, unable to undergo thoracic surgery, or refusing to surgery (according to the eighth edition of TNM staging);
6. Patients with measurable target lesions according to the RECIST 1.1 standard;
7. Patients have not received prior treatment for their NSCLC, including radiotherapy, chemotherapy, surgery and target drugs;
8. Can provide tumor tissue;
9. Adequate organ and marrow function;
10. Fertile female were required to have a serum or urine pregnancy test within 72 hours before the start dose of study medication and the result has been negative;If female of childbearing potential, is willing to use adequate contraception for the course of the study through 90 days after the last dose of study medication; if male with a female partner(s) of child-bearing potential, must agree to use adequate contraception starting with the first dose of study medication through 90 days after the last dose of study medication;
11. Provision of signed ICF.

Exclusion Criteria:

1. Known any distance metastases;
2. Patients with known EGFR gene mutation or ALK fusion mutation;
3. Patients with any active autoimmune disease or history of autoimmune disease;
4. Patients with innate or acquired immune deficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B, hepatitis C or co-infection with hepatitis B and hepatitis C;
5. Subjects requiring systemic treatment with corticosteroids (> 10 mg / day of prednisone or its equivalent) or other immunosuppressants within 14 days prior to the first administration;
6. Patient must not have received a live, attenuated vaccine within 4 weeks prior to the first administration;
7. Any therapy for NSCLC treatment;
8. Patients with other malignant tumors in the past 5 years;
9. Patients with previous or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiologic pneumonia, drug-induced pneumonia and active pneumonia confirmed by imaging;
10. Patients with cardiac insufficiency;
11. Routine urine test indicated that urine protein was >= (+ +), or 24-hour urine protein was >= 1g, or severe liver and kidney dysfunction;
12. Patients with severe infection or fever of unknown origin >38.5 ℃ within 4 weeks prior to the first administration;
13. Patients with known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
14. Pregnant or lactating women; those with fertility who are unwilling or unable to take effective contraceptive measures;
15. Known allergies, hypersensitivity, or intolerance to camrelizumab or its excipients or to pemetrexed or to nab-paclitaxel;
16. Any condition that, in the opinion of the investigator, would interfere with evaluation of the study drug or interpretation of patient safety or study results，or the patient is unlikely to comply with study procedures, restrictions, and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | up to approximately 3 years
  PFS is determined by the Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1).

SECONDARY OUTCOMES:
Overall Survival (OS) | up to approximately 5 years
  OS is defined as the first date of treatment to date of death from any causes.
Objective response rate (ORR) | up to approximately 1 years
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 by investigator.
Disease Control Rate (DCR) | up to approximately 3 years
  DCR is defined as the percentage of patients who have achieved complete response and partial response per RECIST 1.1 by investigator..
Adverse Events (AEs) | up to 18 months
  The number of participants experiencing an AE will be assessed.
PFS at 12 months (PFS12) | up to maximum 12 months
  PFS will be calculated using Kaplan-Meier product limit methods.
PFS at 24 months (PFS24) | up to maximum 24 months
  PFS will be calculated using Kaplan-Meier product limit methods.
PFS at 5 years | up to maximum 5 years
  PFS will be calculated using Kaplan-Meier product limit methods.
OS at 12 months (OS12) | up to maximum 12 months
  OS will be calculated using Kaplan-Meier product limit methods.
OS at 24 months (OS24) | up to maximum 24 months
  OS will be calculated using Kaplan-Meier product limit methods.
OS at 5 years | up to maximum 5 years
  OS will be calculated using Kaplan-Meier product limit methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China